CLINICAL TRIAL: NCT05321927
Title: Transcutaneous Electrical Nerve Stimulation in Persons With MS
Brief Title: TENS in Persons With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-STIM
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcutaneous Electric Nerve Stimulation; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (Sham Comparator): Sham stimulation will be applied over quadriceps femoris and biceps brachii on both sides for 10 min to each muscle group, one at a time. Stimulation is delivered for 10 min to each muscle group, in three 10 minute sessions per week, for 4 weeks.
  Interventions: Device: Sham stimulation
- Strength-training group (Active Comparator): Three training sessions for 10 minutes per muscle group per week, for 4 weeks during which sham stimulation will be applied.
  Interventions: Other: Strength training; Device: Sham stimulation
- Trancutaneous Electrical Nerve Stimulation (TENS) (Active Comparator): Trancutaneous Electrical Nerve Stimulation (TENS) stimulation applied quadriceps femoris and biceps brachii on both sides for 10 min to each muscle group, one at a time. Stimulation is delivered for 10 min to each muscle group, in three 10 minute sessions per week, for 4 weeks.
  Interventions: Device: Trancutaneous Electrical Nerve Stimulation
- TENS with strength training (Experimental): Three training sessions for 10 minutes per target muscle group per week, for 4 weeks during which Trancutaneous Electrical Nerve Stimulation (TENS) stimulation is applied quadriceps femoris and biceps brachii on both sides.
  Interventions: Device: Trancutaneous Electrical Nerve Stimulation; Other: Strength training

INTERVENTIONS:
Device: Trancutaneous Electrical Nerve Stimulation — Transcutaneous Electrical Nerve Stimulation produces an electrical current to stimulate the nerves for therapeutic purposes. continuous high frequency (≥ 50 Hz) stimulation for 5 minutes followed by high frequency (≥ 50 Hz) bursts with 7 pulses per burst for the last 5 minutes.
  Other Names: TENS
  Arms: TENS with strength training; Trancutaneous Electrical Nerve Stimulation (TENS)
Other: Strength training — Three training sessions for 10 minutes per muscle, per week, for four weeks in total.
  Arms: Strength-training group; TENS with strength training
Device: Sham stimulation — Continuous stimulation at 1 Hz for 2 seconds, then no stimulation for 10 seconds. This will alternate for 10 minutes. The intensity equals the intensity that is just felt by the individual.
  Arms: Control group; Strength-training group

SUMMARY:
Persons with multiple sclerosis (pwMS) often have an increased sense of fatigue. Furthermore, they present walking difficulties which negatively affects their mobility and results in an additional increase of fatigue. Previous literature suggests that transcutaneous electrical nerve stimulation (TENS) of leg muscles might increase their walking capacity and decrease perception of fatigue. In the present study we aim to investigate whether TENS of leg muscles reduces walking difficulties and sense of fatigue in pwMS in comparison with a short strength training protocol or no training. A similar aim is addressed after TENS of elbow flexor muscles.

Subjects with relapsing remitting or progressive MS, will undergo transcutaneous electrical nerve stimulation (TENS), strength exercises (SExerc), both TENS and SExerc (COMB) simultaneously, or sham stimulation without training (CON) of both leg and arm muscles. Force and fatigue measurements are performed before, directly after and three weeks after the training sessions and contain walking, fatigue, and strength assessments.

Main study parameters are changes in the scores of i) the six-minute walking test (6-MWT), ii) the perceived walking disability (MSWS-12) and iii) fatigue questionnaires (FSS and MFIS). Additional study parameters are changes in muscle force and muscle fatigability.

ELIGIBILITY:
Inclusion Criteria:

* EDSS score < 7
* MSWS score > 30
* FSS score > 4 or MFIS score > 38.
* no known cardiovascular disorder or having a positive advice on a sport medical examination

Exclusion Criteria:

* being a participant in an exercise study
* having a psychiatric disorder
* having cognitive or communication problems which reduces the capacity to understand instructions
* planned a change in medication during the training period
* having a neurological disorder other than MS
* having cardiovascular disorders and no positive advice from a sport medical examination
* having a pacemaker or another implantable electronic apparatus.
* being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 6 weeks
  This test assesses submaximal aerobic capactity. Subjects walk for 6 minutes starting at mark on the floor at the beginning of a 30-m long hallway and walk to the next mark at the end of the hallway as quickly as possible, but safely. The distance which is walked by the subject is measured. Subjects may use assistive devices when performing the task.
chair-stand test | 6 weeks
  This test assesses functional lower extremity strength. Subjects sit on a chair and stand up repeatedly for 30 s. Arms of the subject are crossed and held against the chest. The number of cycles of standing up from sitting are counted.
Fatigue Severity Scale (FSS) | 6 weeks
  This is a questionnaire related to the impact of fatigue on daily life. The questionnaire consists of 9 questions with a 7-point scale ranging from 'completely agree' to 'completely disagree'. The total score ranges from 9 to 63; higher scores reflect a higher impact.
Modified Fatigue Impact Scale (MFIS) | 6 weeks
  This is a questionnaire related to sense of fatigue. The questionnaire consist of 21 questions providing assessment of the effect of fatigue in terms of physical, cognitive and psychosocial function. The total score ranges from 0 to 84; higher scores reflect a higher impact of fatigue.
12-item MS walking scale (MSWS-12) | 6 weeks
  This is a patient-base measure of walking ability. The questionnaire consists of 12 items with a 5-point scale ranging from 'not at all' to 'extremely'. The total score ranges from 5 to 60, with higher scores reflecting more walking difficulties.

SECONDARY OUTCOMES:
Elbow flexor muscle force (maximal and submaximal levels) | 6 weeks
  Maximal voluntary force (MVC) of the elbow flexors is measured with a custom-built dynamometer. Subjects are seated in a chair with their arm abducted and in 90° of flexion with their non-dominant arm strapped to the force transducer. Subjects are instructed to contract their elbow flexors as rapidly and forcefully as possible and to maintain force generation for 5 s. MVC is determined as the peak force.
Knee extensor muscle force (maximal and submaximal levels) | 6 weeks
  Maximal voluntary force (MVC) of the knee extensors is measured with a custom-built dynamometer. Subjects are seated in a chair with the knee and hip in 90° of flexion with their non-dominant lower leg strapped to the chair's lever arm (~ 10 cm up to lateral malleolus). Subjects are instructed to contract their knee extensors as rapidly and forcefully as possible and to maintain force generation for 5 s. MVC is determined as the peak force.
Handgrip force | 6 weeks
  Maximal voluntary force (MVC) of the handgrip is measured with a hydraulic hand dynamometer (JAMAR Hand Dynamometer). The measurement is repeated 3 times and averaged.
Effort during submaximal contractions with elbow flexors | 6 weeks
  Subjects are asked to produce different submaximal force levels of the elbow flexors (20, 30, 50 and 70%) and rate their perceived effort (scale 1-10) that was needed to generate this force level.
Effort during submaximal contractions with knee extensors | 6 weeks
  Subjects are asked to produce different submaximal force levels of the knee extensors (20, 30, 50 and 70%) and rate their perceived effort (scale 1-10) that was needed to generate this force level.

OTHER OUTCOMES:
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | 6 weeks
  A self-report questionnaire with 54 items used to quantify health-related quality of life. Generates two separate composite scores for physical and mental health (0-100); higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Inge CAT Zijdewind, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No